CLINICAL TRIAL: NCT07309978
Title: Assessment Of Difficult Airway Predictors: A Prospective Comparison Of Upper Airway Ultrasound And Conventional Anthropometric Measures
Status: Not yet recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Sami Eksert, anesthesiology specialist, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Other Study IDs: AEŞH-EK-2-25-276
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Prediction of Difficult Airway; Difficult Airway Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Cohort: This cohort includes all adult participants undergoing airway evaluation with upper airway ultrasound and standard anthropometric measurements. No interventions are applied; participants are observed prospectively to assess the predictive value of ultrasound parameters for difficult airway.

SUMMARY:
This prospective observational study aims to evaluate whether upper airway ultrasound measurements can improve the prediction of difficult airway compared with conventional anthropometric assessments. Adult patients undergoing elective procedures requiring airway management will be included. Ultrasound parameters such as tongue thickness, anterior neck soft tissue thickness, and hyomental distance will be measured before airway intervention. Standard clinical predictors (Mallampati score, thyromental distance, neck circumference, etc.) will also be recorded. The primary objective is to determine the diagnostic accuracy of ultrasound-based measurements in predicting difficult laryngoscopy and intubation. The study seeks to provide evidence supporting the integration of upper airway ultrasound into routine pre-anesthetic airway evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-99 years
* Patients scheduled for elective surgery under general anesthesia
* ASA Physical Status I-III
* Able to provide informed consent
* Undergoing preoperative airway evaluation

Exclusion Criteria:

* - Emergency surgery cases
* Age <18 years
* ASA Physical Status IV-V
* Pregnant or breastfeeding patients
* Patients with limited cooperation or inability to provide consent
* Known anatomical airway anomalies or previous major neck surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (18-99 years) scheduled for elective surgery under general anesthesia at a tertiary care hospital. Participants represent typical surgical patients requiring preoperative airway assessment. No healthy volunteers will be enrolled. Only ASA I-III patients who can provide informed consent will be included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-07-25 (Estimated); Study Completion 2027-12-25 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of ultrasound airway measurements for predicting difficult mask ventilation | Preoperative assessment (within 1 hour before induction of anesthesia)
  Evaluation of the sensitivity, specificity, and area under the ROC curve (AUC) of ultrasound-based airway measurements-tongue thickness, hyoid-to-skin distance, and epiglottis-to-skin distance-in predicting difficult mask ventilation. These ultrasound parameters will be compared with conventional anthropometric airway assessment tests to determine their predictive performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rastogi A, Singh AK, Srivastava D, Kannaujia AK, Singh TK, Mishra P. Evaluation of ultrasound measured tongue thickness, tongue thickness-thyromental distance ratio, and skin-to-epiglottis distance in predicting unanticipated difficult laryngoscopy. J Anaesthesiol Clin Pharmacol. 2025 Jan-Mar;41(1):151-157. doi: 10.4103/joacp.joacp_423_23. Epub 2025 Jan 23. PMID 40026745
- [Background] Yao W, Wang B. Can tongue thickness measured by ultrasonography predict difficult tracheal intubation? Br J Anaesth. 2017 Apr 1;118(4):601-609. doi: 10.1093/bja/aex051. PMID 28403413
- [Background] Roth D, Pace NL, Lee A, Hovhannisyan K, Warenits AM, Arrich J, Herkner H. Airway physical examination tests for detection of difficult airway management in apparently normal adult patients. Cochrane Database Syst Rev. 2018 May 15;5(5):CD008874. doi: 10.1002/14651858.CD008874.pub2. PMID 29761867